CLINICAL TRIAL: NCT06055270
Title: Stellate Ganglion Block with Lidocaine for the Treatment of COVID-19-Induced Parosmia: Double-Blinded, Placebo-Controlled Randomized Clinical Trial
Brief Title: Stellate Ganglion Block with Lidocaine for the Treatment of COVID-19-Induced Parosmia
Acronym: Stella
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, Leigh Sowerby, MD, MHM, FRCSC Associate Professor, Rhinology and Anterior Skull Base Surgery, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ReDA 13983
Record Dates: First submitted 2023-09-22; First posted 2023-09-26 (Actual); Last update posted 2024-10-23 (Actual); Status verified 2024-04

CONDITIONS: Parosmia
Keywords: Long-COVID; Olfactory disfunction; smell; olfaction; anosmia; bad smell
MeSH Terms: conditions — Olfaction Disorders; Post-Acute COVID-19 Syndrome; Anosmia | interventions — Autonomic Nerve Block

STUDY DESIGN:
Intervention Model Description: Double-Blinded, Placebo-Controlled Randomized Clinical Trial
Who Masked: Participant, Investigator
Masking Description: Study statistician
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo Group (Placebo Comparator): The placebo sham injection will be performed in an identical fashion as the stellate ganglion block, with the exception of using 8 mL of 0.9% saline injection instead of Lidocaine.
  Interventions: Other: Placebo
- Stellate Ganglion Block (Experimental): The ultrasound-guided stellate ganglion blocks will be performed by a pain management specialist with extensive experience performing these blocks. The first SGB at the initial visit will be performed on the right side, and the second SGB will be on the left side 5-10 days after the first SGB, given that the patient tolerated the first SGB.
  Interventions: Procedure: Stellate Ganglion Block

INTERVENTIONS:
Procedure: Stellate Ganglion Block — All SGBs will be performed by a board-certified anesthesiologist and pain management specialist with extensive experience performing SGBs. The laterality of the SGB will be randomized between the left and right sides of the neck. Participants will be asked to abstain from eating and drinking for 8 hours prior to the SGB. Using ultrasound guidance, the transverse process of the C6 vertebra is identified. Color-doppler is used to identify blood vessels. A 27-gauge needle is used to anesthetize the superficial skin with 1% lidocaine. Then, a 21-gauge ultrasound needle is advanced using an in-plane technique from lateral to medial with careful avoidance of neurovascular structures. After negative aspiration, 8 mL of 1% Lidocaine is deposited beneath the prevertebral fascia and above the Longus coli muscle into the stellate ganglion.
  Other Names: SGB; sympathetic block
  Arms: Stellate Ganglion Block
Other: Placebo — The placebo sham injection will be performed in an identical fashion as the stellate ganglion block, with the exception of using 8 mL of 0.9% saline injection instead of Lidocaine
  Other Names: Placebo sham injection
  Arms: Placebo Group

SUMMARY:
Chronic olfactory dysfunction, both hyposmia and parosmia, from the COVID-19 pandemic is a growing public health crisis, affecting up to 1.2 million people in the United States. Olfactory dysfunction significantly impacts one's quality of life by decreasing the enjoyment of foods, creating environmental safety concerns, and affecting one's ability to perform specific jobs. Olfactory loss is also an independent predictor of anxiety, depression, and mortality.

Recent research suggests that parosmia, more so than hyposmia, can increase anxiety, depression, and even suicidal ideation. While the pandemic has advanced the scientific community's interest in combating the burgeoning health crisis, few effective treatments currently exist for olfactory dysfunction. Persistent symptoms after an acute COVID-19 infection, or "Long COVID" symptoms, have been hypothesized to result from sympathetic nervous system dysfunction. Stellate ganglion blocks have been proposed to treat this hyper-sympathetic activation by blocking the sympathetic neuronal firing and resetting the balance of the autonomic nervous system. Studies before the COVID-19 pandemic have supported a beneficial effect of stellate ganglion blocks on olfactory dysfunction, and recent news reports and a published case series have described a dramatic benefit in both olfactory function and other long COVID symptoms in patients receiving stellate ganglion blocks. A previous pilot study using stellate ganglion blocks of 20 participants with persistent COVID-19 olfactory dysfunction resulted in modest improvements in subjective olfactory function, smell identification, and olfactory-specific quality of life, but it lacked a control group.

Therefore, we propose a double-blinded, placebo-controlled, randomized clinical trial assessing the efficacy of a stellate ganglion block with Lidocaine versus saline injection in up to 50 participants with persistent COVID-19-associated olfactory dysfunction.

DETAILED DESCRIPTION:
This will be a double-blinded, placebo-controlled, randomized clinical to assess the efficacy of Stellate Ganglion Block with Lidocaine 1% (8mL). Participants with parosmia will be randomly assigned to SGB with Lidocaine 1% (8mL) or Placebo (saline solution). Baseline assessment will happen in person and will consist on demographic information, Parosmia Olfactory Dysfunction Outcomes Rating (DisODOR), Clinical Global Impression: Severity Scale (CGI-S), University of Pennsylvania Smell Identification Test (UPSIT), Long-COVID Questionnaire (LCQ), Olfaction Catastrophizing Scale (OCS), Hospital Anxiety and Depression Scale (HADS), Pre-Intervention Expectations. Then, after the assigned interventional procedures are performed three remote visits will be performed as follow-ups (1, 3, and 12 months), in which the variables above will be reassessed.

ELIGIBILITY:
Inclusion Criteria:

1. Adults age 18 to 70
2. Diagnosis of COVID-19 at least 6 months prior to study enrollment with self-reported parosmia
3. Ability to read, write, and understand English
4. Score of at least 15 on DiSODOR

Exclusion Criteria:

1. History of smell loss or change prior to COVID-19 infection
2. History of conditions known to impact olfactory function:

   1. Chronic rhinosinusitis
   2. History of prior sinonasal or skull base surgery
   3. Neurodegenerative disorders (Parkinson's disease, Huntington's disease, Amyotrophic lateral sclerosis, Lewy body dementia, frontotemporal dementia)
3. Currently using concomitant therapies specifically for the treatment of olfactory dysfunction
4. Inability to tolerate a needle injection into the neck
5. History of coexisting conditions that make SGB contraindicated:

   1. Unilateral vocal cord paralysis
   2. Severe chronic obstructive pulmonary disease (FEV1 between 30-50% of predicted)
   3. Recent myocardial infarction within the last year
   4. Glaucoma
   5. Cardiac conduction block of any degree
6. Currently taking blood thinners or antiplatelet agents
7. Allergy to local anesthetic
8. Inability to extend the neck for any reason (e.g., severe arthritis)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2024-02-15 (Actual); Primary Completion 2025-12-24 (Estimated); Study Completion 2026-05-15 (Estimated)

PRIMARY OUTCOMES:
Parosmia Olfactory Dysfunction Outcomes Rating (DisODOR) | Baseline, 1, 3, and 12 months after SGB
  The DisODOR is a disease-specific questionnaire that assesses for physical problems, functional limitations, and emotional consequences of parosmia secondary to any etiology. The instrument contains 29 total items with each scored on a 5-point Likert scale from 0 to 4. The minimal clinically important difference (MCID) for the instrument is 15.

SECONDARY OUTCOMES:
Clinical Global Impression - Severity Scale (CGI-S) | Baseline
  The baseline severity of parosmia will be measured with the CGI-S scale. The CGI-S scale measures disease severity in clinical condition based on a 5-point Likert scale.
Clinical Global Impression - Improvement Scale (CGI-I) | 1, 3, and 12 months after SGB
  The overall response to treatment will be measured with the CGI-I scale. The CGI-I Scale measures response to treatment for a number of disorders and has good internal consistency and validity.32 The CGI-I scale measures change in clinical condition based on a 7-point Likert scale. The CGI-I for parosmia asks, "Compared to before your stellate ganglion block, how would you describe your parosmia (things do not smell the same as you remember)?" Response options for each are: (1) Much better now than before, (2) Moderately better now than before, (3) Slightly better now than before, (4) About the same, (5) Slightly worse now than before, (6) Moderately worse now than before, and (7) Much worse now than before. Responders are defined as those who report "slightly better now than before" or greater.
University of Pennsylvania Smell Identification Test (UPSIT, Sensonics, New Jersey). | Baseline
  The UPSIT is a test of olfactory identification and consists of four 10-page booklets, with a total of 40 items. On each page, there is a different "scratch and sniff" strip and four choice options. Subjects are asked to scratch each strip with a pencil to release the scents, detect the smell, and identify the smell from the four choice options. The UPSIT comes from a scoring rubric that identifies the normalcy benchmark based on age and gender, which is >34 in women and >33 in men.33,34 The UPSIT is commercially available, takes 10-15 minutes to complete, and is the gold standard test to assess smell identification. The minimal clinically important difference of the UPSIT is 4.
Long-COVID Questionnaire (LCQ) | Baseline, 1, 3, and 12 months after SGB
  Symptoms assessed via the LCQ are derived from the Symptom Burden Questionnaire for Long Covid35, which included tiredness/fatigue, shortness of breath, brain fogginess, headache, cough, depression, low-grade fevers, palpitations, dizziness, muscle pain, and joint pains. At baseline, participants are asked to rank the current severity of each problem on a 5-point Likert scale. At each follow-up visit, participants are asked to rank their overall improvement in each of the 11 symptoms compared to their symptoms prior to their first SGB. The improvement options are based on the CGI-I 7-point Likert scale.
Olfaction Catastrophizing Scale (OCS) | Baseline, 1, 3, and 12 months after SGB
  The pain catastrophizing scale (PCS) was developed to measure the negative mental response to actual or anticipated pain. The OCS was derived from the validated PCS to similarly measure the negative mental response to smell dysfunction loss. Multiple thoughts/feelings will be assessed on a 5-point Likert scale with a maximum score of 52. At each visit, subjects will be asked to complete the OCS.
Hospital Anxiety and Depression Scale (HADS) | Baseline, 1, 3, and 12 months after SGB
  The HADS was developed for screen for anxiety and depression in the general population. It consists of 7 questions for anxiety and 7 questions for depression each ranked on a 4-point Likert Scale. A score of 0-7 is considered normal, 8-10 is borderline abnormal anxiety or depression, and a score of 11-21 corresponds with screening positive for anxiety or depression. Subjects will be screened for anxiety and depression on their initial visit.
Pre-Intervention Expectations | Baseline
  A significant number of social media and news stories have discussed anecdotal success of stellate ganglion blocks for COVID-19-induced olfactory dysfunction. As a result, we propose that participants may have a distorted pre-operative expectation that may affect their subjective rating of improvement in olfaction. Therefore, participants will be asked at baseline, "How confident are you that the stellate ganglion block will improve your smell loss or smell distortion?" Possible answer choices: Not at all, Slightly confident, Somewhat confident, Very confident, Extremely confident.
Patient Satisfaction with Treatment | 1, 3, and 12 months after SGB
  Participants will be asked at the 1-month virtual visit, "Overall, how satisfied were you with the stellate ganglion block treatment for your parosmia?" Possible answer choices: 1) Completely dissatisfied, 2) Mostly dissatisfied, 3) Somewhat dissatisfied, 4) Neither satisfied or dissatisfied, 5) Somewhat satisfied, 6) Mostly satisfied, 7) Completely satisfied. Patients will also be asked at the final visit, "Would you recommend this treatment to a family member or close friend who also suffers from chronic smell loss due to COVID-19?" Possible answer choices: 1) Yes, 2) No.
Assessment of the Blind | 1 Month after SGB
  Immediately after the initial injection, participants will be asked, "Which intervention do you think you received?" Answer choices: 1)Lidocaine (active medication) 2) Saline (placebo).

CONTACTS AND LOCATIONS:
Locations (1):
- St. Joseph's Hospital London, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hintschich CA, Fischer R, Hummel T, Wenzel JJ, Bohr C, Vielsmeier V. Persisting olfactory dysfunction in post-COVID-19 is associated with gustatory impairment: Results from chemosensitive testing eight months after the acute infection. PLoS One. 2022 Mar 23;17(3):e0265686. doi: 10.1371/journal.pone.0265686. eCollection 2022. PMID 35320821
- [Background] Fortunato F, Martinelli D, Iannelli G, Milazzo M, Farina U, Di Matteo G, De Nittis R, Ascatigno L, Cassano M, Lopalco PL, Prato R. Self-reported olfactory and gustatory dysfunctions in COVID-19 patients: a 1-year follow-up study in Foggia district, Italy. BMC Infect Dis. 2022 Jan 22;22(1):77. doi: 10.1186/s12879-022-07052-8. PMID 35065619
- [Background] Khan AM, Kallogjeri D, Piccirillo JF. Growing Public Health Concern of COVID-19 Chronic Olfactory Dysfunction. JAMA Otolaryngol Head Neck Surg. 2022 Jan 1;148(1):81-82. doi: 10.1001/jamaoto.2021.3379. PMID 34792577
- [Background] Lerner DK, Garvey KL, Arrighi-Allisan AE, Filimonov A, Filip P, Shah J, Tweel B, Del Signore A, Schaberg M, Colley P, Govindaraj S, Iloreta AM. Clinical Features of Parosmia Associated With COVID-19 Infection. Laryngoscope. 2022 Mar;132(3):633-639. doi: 10.1002/lary.29982. Epub 2021 Dec 13. PMID 34870334
- [Background] Schambeck SE, Crowell CS, Wagner KI, D'Ippolito E, Burrell T, Mijocevic H, Protzer U, Busch DH, Gerhard M, Poppert H, Beyer H. Phantosmia, Parosmia, and Dysgeusia Are Prolonged and Late-Onset Symptoms of COVID-19. J Clin Med. 2021 Nov 12;10(22):5266. doi: 10.3390/jcm10225266. PMID 34830550
- [Background] Hopkins C, Surda P, Vaira LA, Lechien JR, Safarian M, Saussez S, Kumar N. Six month follow-up of self-reported loss of smell during the COVID-19 pandemic. Rhinology. 2021 Feb 1;59(1):26-31. doi: 10.4193/Rhin20.544. PMID 33320115
- [Background] Keller A, Malaspina D. Hidden consequences of olfactory dysfunction: a patient report series. BMC Ear Nose Throat Disord. 2013 Jul 23;13(1):8. doi: 10.1186/1472-6815-13-8. PMID 23875929
- [Background] Santos DV, Reiter ER, DiNardo LJ, Costanzo RM. Hazardous events associated with impaired olfactory function. Arch Otolaryngol Head Neck Surg. 2004 Mar;130(3):317-9. doi: 10.1001/archotol.130.3.317. PMID 15023839
- [Background] Pang NY, Song HJJMD, Tan BKJ, Tan JX, Chen ASR, See A, Xu S, Charn TC, Teo NWY. Association of Olfactory Impairment With All-Cause Mortality: A Systematic Review and Meta-analysis. JAMA Otolaryngol Head Neck Surg. 2022 May 1;148(5):436-445. doi: 10.1001/jamaoto.2022.0263. PMID 35389456
- [Background] Addison AB, Wong B, Ahmed T, Macchi A, Konstantinidis I, Huart C, Frasnelli J, Fjaeldstad AW, Ramakrishnan VR, Rombaux P, Whitcroft KL, Holbrook EH, Poletti SC, Hsieh JW, Landis BN, Boardman J, Welge-Lussen A, Maru D, Hummel T, Philpott CM. Clinical Olfactory Working Group consensus statement on the treatment of postinfectious olfactory dysfunction. J Allergy Clin Immunol. 2021 May;147(5):1704-1719. doi: 10.1016/j.jaci.2020.12.641. Epub 2021 Jan 13. PMID 33453291